CLINICAL TRIAL: NCT05249881
Title: "Efficacy of Once-weekly GLP 1 Analogue: Semaglutide. A Multicenter Experience From Pakistan."
Brief Title: "Efficacy of Once Weekly GLP 1 Analogue: Semaglutide. A Multicenter Experience From Pakistan."
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Rehman Medical Institute - RMI (Other)
Responsible Party: Principal Investigator, NASEER AHMED, Assistant Professor, Aga Khan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 07125
Record Dates: First submitted 2022-02-09; First posted 2022-02-22 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2; Weight Change, Body
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Body Weight Changes | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- semaglutide (Other): semaglutide is an anti-diabetic medication used for the treatment of type 2 diabetes and long-term weight management. Semaglutide acts like human glucagon-like peptide-1 in that it increases insulin secretion, thereby increasing sugar metabolism
  Interventions: Drug: Semaglutide Pen Injector

INTERVENTIONS:
Drug: Semaglutide Pen Injector — All Diabetes mellitus type2 patients fulfilling the inclusion criteria, will receive 0.25mg Semaglutide injection per week and after two weeks dosage will be escalated to 0.5 mg/week for next 10 weeks.
  Other Names: Ozempic

SUMMARY:
A prospective interventional trial for 9 months will be carried out on 300 type-2 diabetes mellitus volunteer patients who are above 18-year-old and participants will be selected through consecutive sampling and will be evaluated on the basis of glycemic index and history of patients. Selected parameters will be measured at baseline and after the 12 weeks of therapy. Statistical analysis will be carried out by SPSS, ANOVA, and t-test.

From this experimental design, we are expecting improvement in the management of glycemic index, reduction in systolic and diastolic blood pressure, and reduction in weight GLP-1 naive patients.

DETAILED DESCRIPTION:
Patients will be recruited from all the 12 centers included in the trial across Pakistan and data will be electronically transferred to the main center. All GLP-1 naive patients fulfilling the inclusion criteria will be recruited after informed written consent and started on Semaglutide injection 0.25mg for 2 weeks and will be escalated to 0.5 mg for the next 10 weeks. Socio-Demographic Data and health vitals including height, weight, BMI, baseline HbA1c, FBS and RBS will be recorded in preset Performa. All those who agree to participate will be given structured education on diet and exercise and those willing to comply will be recruited. A research assistant will be recruited and trained to teach the injection technique and discuss the adverse effects of Semaglutide to the participants. Patients taking DPP-4 inhibitors will be switched to GLP-1 analogue and only a single drug change in the form of adding Semaglutide will be done at the time. Semaglutide injection technique will be explained to the patient and one injection at a time will be provided to the patient to ensure compliance and avoid bias in the study. Patients will be asked to revisit after 4 weeks with the used injection device. After completion of 3 months of treatment vitals including height, weight, BMI, baseline HbA1c, FBS and RBS will be recorded in preset Performa.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female Type 2 Diabetic patients with age ≥18 years.
* Patients with HbA1c ≥ 7.5 % - ≤ 10.0%
* Patients with BMI ≥ 30

Exclusion Criteria:

* Patients with Type 1 Diabetes Mellitus
* Patients with Gestational Diabetes Mellitus.
* Patients with Chronic Renal Failure with eGFR of ≤ 30ml/min
* Patient already on another GLP 1 analogue
* The patient stopped any GLP1 analogue treatment less than 3 months back.
* Patients with history of chronic pancreatitis or pancreatic cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in glycemic Index in Diabetes mellitus type-2 Patients | 3 months
  Once weekly Semaglutide may result to remarkably change HbA1c level with in 3 months of use

SECONDARY OUTCOMES:
Weight Changes in Obese People | 3 months
  use of semaglutide may help obese people in controlling their weight gain.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Rehman Medical Institute, Peshawar, KPK
  - Aga Khan University, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No